CLINICAL TRIAL: NCT01865968
Title: Phase IV Trial to Compare the Safety, Immunogenicity,Three-year Immune Persistence of Inactivated Hepatitis A Vaccine (HAV) With One- or Two-dose Regimen and Live Attenuated HAV With One-dose Regimen in Chinese Young Adults, and to Evaluate the Immunogenicity of a Booster Dose.
Brief Title: Comparison of Immunogenicity and Safety of Inactivated and Live Attenuated Hepatitis A Vaccines in Young Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRO-HA-4009
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Hepatitis A
Keywords: inactivated HAV vaccine; live attenuated HAV vaccine; immunogenicity; safety
MeSH Terms: conditions — Hepatitis A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Inactivated HAV vaccine (Experimental): Healthy undergraduate students aged 16 to 25 years with anti-HAV negative received inactivated HAV vaccine containing 500u/vial with one-dose regimen.
  Interventions: Biological: Inactivated HAV vaccine
- Live attenuated HAV vaccine (Active Comparator): Healthy undergraduate students aged 16 to 25 years with anti-HAV negative received live attenuated HAV vaccine containing 6.50 lgCCID50/vial with one-dose regimen.
  Interventions: Biological: Live attenuated HAV vaccine
- Two-dose inactivated HAV vaccine (Experimental): Healthy undergraduate students aged 16 to 25 years with anti-HAV negative received inactivated HAV vaccine containing 500u/vial with two-dose regimen.
  Interventions: Biological: Inactivated HAV vaccine

INTERVENTIONS:
Biological: Inactivated HAV vaccine — Hepatitis A vaccine (Healive), 500 u per dose per 0.5 millilitre. Vaccines will be administered with one-dose or two-dose regimen of the arm 6 months apart in the deltoid muscle.
  Other Names: Inactivated hepatitis A vaccines
  Arms: Inactivated HAV vaccine; Two-dose inactivated HAV vaccine
Biological: Live attenuated HAV vaccine — Live attenuated hepatitis A vaccine, 6.50 lgCCID50 per dose per 0.5 millilitre. Vaccines will be administered with one-dose regimen in the deltoid muscle.
  Other Names: Live attenuated hepatitis A vaccines
  Arms: Live attenuated HAV vaccine

SUMMARY:
A phase IV, randomization, single center, controlled clinical trial to compare the safety, immunogenicity,three-year immune persistence of inactivated hepatitis A vaccine (HAV) with one- or two-dose regimen and live attenuated HAV with one-dose regimen in Chinese young adults, and to evaluate the immunogenicity of a booster dose.

DETAILED DESCRIPTION:
Healthy undergraduate students aged 16 to 25 years with anti-HAV negative were randomly divided into three groups. Group A and B were administrated with one-dose inactivated and live attenuated hepatitis A vaccines respectively; Group C was immunized with two doses of an inactivated vaccine with 6 months apart. Blood samples were collected at month 1, and 12, 24 and 36 for anti-HAV titers determination. Safety observation in 30 minutes' duration after vaccinations and injection-site reactions and systemic reactions for three consecutive days were recorded to assess the safety of investigational vaccines. At Month 36, subjects who received one dose of inactivated or live attenuated HAV were administrated a booster dose and then were taken blood samples one month later for anti-HAV titers determination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy undergraduate students aged 16 to 25 years
* Sign the informed consent
* Provide ID

Exclusion Criteria:

* Axillary temperature > 37.0 centigrade at the time of dosing
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine
* Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
* Autoimmune disease or immunodeficiency
* Congenital malformation, developmental disorders or serious chronic diseases (such as Down's syndrome, diabetes, sickle cell anemia or neurological disorders)
* Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM injections or blood draws
* History or family history of convulsions, epilepsy, brain disease and psychiatric
* History of any blood products within 3 months
* Administration of any other investigational research agents within 30 days
* Administration of any live attenuated vaccine within 30 days
* Administration of subunit or inactivated vaccines within 14 days
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent
* anti-HBsAg positive
* anti-HAV positive
* Pregnancy test result is positive

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 239 (Actual)
Dates: Start 2008-10; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
concentration of antibody to hepatitis A virus | 37 months
  Anti-HAV antibody geometric mean concentrations pre-vaccination, and at month 1, and 12, 24 and 36, and 1 months (month 37) after the booster vaccination.

SECONDARY OUTCOMES:
reported side effects and adverse events | 37 months
  After each dose, solicited injection-site and general adverse events (AEs) were recorded for 7 days and unsolicited AEs were recorded for 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhuang, Ph.D, MD, Principal Investigator — Medical school of Peking University
Locations (1):
- Nanchang Center for Disease prevention and Control, Nanchang, Jiangxi, China

REFERENCES:
- [Derived] Liu XE, Chen HY, Liao Z, Zhou Y, Wen H, Peng S, Liu Y, Li R, Li J, Zhuang H. Comparison of Immunogenicity Between Inactivated and Live Attenuated Hepatitis A Vaccines Among Young Adults: A 3-Year Follow-up Study. J Infect Dis. 2015 Oct 15;212(8):1232-6. doi: 10.1093/infdis/jiv213. Epub 2015 May 12. PMID 25969561